CLINICAL TRIAL: NCT06393673
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2 Study to Investigate the Efficacy and Safety of HS-10384 in Postmenopausal Women Suffering From Vasomotor Symptoms (Hot Flashes)
Brief Title: A Study to Find the Best Dose of HS-10384 to Treat Vasomotor Symptoms in Postmenopausal Women
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10384-201
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Vasomotor Symptoms
Keywords: HS-10384; Vasomotor symptoms; postmenopausal women

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HS-10384 Dose 1 (Experimental): Dose level 1 of HS-10384
  Interventions: Drug: HS-10384 tablet Dose 1; Drug: HS-10384-matched placebo tablets
- HS-10384 Dose 2 (Experimental): Dose level 2 of HS-10384
  Interventions: Drug: HS-10384 tablet Dose 2; Drug: HS-10384-matched placebo tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: HS-10384-matched placebo tablets

INTERVENTIONS:
Drug: HS-10384 tablet Dose 1 — Administered orally QD
  Arms: HS-10384 Dose 1
Drug: HS-10384 tablet Dose 2 — Administered orally QD
  Arms: HS-10384 Dose 2
Drug: HS-10384-matched placebo tablets — Administered orally QD

SUMMARY:
A randomized, double-blind, placebo-controlled phase 2 clinical study to evaluate the efficacy and safety of HS-10384 in postmenopausal women suffering from vasomotor symptoms.

DETAILED DESCRIPTION:
The phase 2 study is consisted with 2 doses. The aim is to detect the efficacy, safety, pharmacokinetics and pharmacodynamics characteristics of HS-10384 in participants with vasomotor symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 40 and 65 years old (including extremes);
2. The body mass index at screening is between 18.5~30 kg/m2 (including extremes)；
3. Subjects are postmenopausal women at screening as qualified by any of the following criteria: spontaneous amenorrhea ≥ 12 months, or spontaneous amenorrhea ≥ 6 months and FSH>40 IU/L (without other obvious pathological or physiological reasonsbefore screening), or documented surgical sterilization (such as hysterectomy, bilateral salpingectomy or bilateral oophorectomy, etc.);
4. At least 50 moderate to severe vasomotor symptoms per week (ie, 7 consecutive days), or 7 moderate to severe vasomotor symptoms per day (ie, 7 consecutive days) recorded in the daily diary during the screening period;
5. The blood pregnancy test of female subjects at baseline period is negative.

Exclusion Criteria:

1. Participants with disease history of unexplained uterine bleeding, endometrial hyperplasia, ovarian tumor, pituitary tumor, or other diseases evaluated by the principal investigator as not suitable for this study;
2. Have a history of migraine within 3 months before screening;
3. Uncontrolled hypertension and a systolic blood pressure ≥140 mmHg and/or a diastolic blood pressure ≥90 mmHg;
4. Previous or current history of a malignant tumor, except for basal cell carcinoma;
5. Participants with clinically significant diseases (such as neuropsychiatric system, cardiovascular system, urinary system, digestive system, respiratory system, skeletal muscle system, endocrine and metabolic system, blood system, skin disease, immune system, tumor, etc.) were evaluated by the researcher as not suitable for this study;
6. Within 4 weeks or 5 half-lives (whichever is longer) before taking drug, participants have taken hormonal treatment, hormonal contraceptive or other therapy due to VMS;
7. Within 4 weeks or 5 half-lives (whichever is longer) before screening, and during the whole study period, it is expected to take any medicine and health care products, including prescription drugs, immunomodulator or Chinese herbal medicine, etc.;
8. Participants have participated in any interventional study or taken study drugs within 3 months before screening;
9. Judged by the Investigator to be unsuited to participate in the study based on findings observed during physical examination, vital sign assessment, or 12-lead electrocardiogram (ECG), et al.;
10. Active liver disease or jaundice, or values of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 x the upper limit of normal (ULN); or total bilirubin or direct bilirubin >1.5 x ULN;
11. Creatinine >1.5 x ULN; or estimated glomerular filtration rate (eGFR) using the CKD-EPI formula ≤59 mL/min/1.73 sqm at the screening visit;

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in the frequency of moderate to severe vasomotor symptoms from baseline to Week 4; | Baseline to Week 4
Mean change in the frequency of moderate to severe vasomotor symptoms from baseline to Week 12; | Baseline to Week 12
Mean change in the severity of moderate to severe vasomotor symptoms from baseline to Week 4; | Baseline to Week 4
Mean change in the severity of moderate to severe vasomotor symptoms from baseline to Week 12. | Baseline to Week 12

SECONDARY OUTCOMES:
Mean change in the frequency of moderate and severe vasomotor symptoms from baseline to each study week; | Baseline to Week 15
Mean change in the severity of moderate and severe vasomotor symptoms from baseline to each study week; | Baseline to Week 15
Mean change in the hot flash score of moderate and severe vasomotor symptoms from baseline to each study week; | Baseline to Week 15
Mean percent reduction of 50% and 100% of moderate and severe vasomotor symptoms from baseline to each study week. | Baseline to Week 15
Incidence and severity of treatment-emergent adverse events; | Baseline to Week 15
Number of participants with clinical laboratory abnormalities; | Baseline to Week 15
Number of participants with abnormalities of vital signs | Baseline to Week 15
Number of participants with abnormalities of physical examinations | Baseline to Week 15
Change from baseline in ECG parameters | Baseline to Week 15
Change from baseline in plasma bone density marker concentrations | Baseline to Week 15
Change from baseline in Endometrial health assessment. | Baseline to Week 15

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences (CAMS)Peking Union Medical College (PUMC), Shanghai, Shanghai Municipality, China